CLINICAL TRIAL: NCT02148497
Title: Viability Study of a Multi-Colored Videokeratoscope With Extended Timescale Data
Brief Title: Multi-Colored Placido Disk Viability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Geunyoung Yoon, Principle Investigator, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 51771
Record Dates: First submitted 2014-04-15; First posted 2014-05-28 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Dry Eye; Sjogren's Disease; Healthy
Keywords: volunteers
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Eye Disease or Sjogren's Disease (Other): Capturing images of the tear surface using the multi-colored Placido disk
  Interventions: Procedure: Multi-colored Placido disk imaging
- Control (Other): Capturing images of the tear surface using the multi-colored Placido disk
  Interventions: Procedure: Multi-colored Placido disk imaging

INTERVENTIONS:
Procedure: Multi-colored Placido disk imaging — The multi-colored Placido disk instrument records the tear surface using video imaging.

SUMMARY:
The purpose of this study is to show that the multi-colored Placido Disk set-up can get reliable data over long time periods.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clinically diagnosed Dry Eye or Sjörgren's syndrome.
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions that are deemed confounding to the data as determined by the PI)
* Ability to give informed consent
* Willing to spend time for the study; approximately 30 minutes for a visit
* Either gender
* Any racial or ethnic origin

Exclusion Criteria:

* Use of any prescription ocular medication (such as but not limited to, glaucoma medications and Restasis) used within 14 days of the screening visit or started prior to the measurement visit(s).
* Current eye disease, infection or inflammation that affects the surface of the eye such as, but not limited to blepharitis and ocular allergy.
* Past eye surgery, such as, but not limited to, refractive surgery. Subjects who have had cataract surgery less than one year ago.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Tear film break-up time | up to 3 seconds
  The multi-colored Placido disk will collect images of the tear film with the aim to have usable data for more extended periods of time. This instrument measures tear film break-up time in seconds using a video recording of the tear surface.

CONTACTS AND LOCATIONS:
Overall Officials: Geunyoung Yoon, PhD, Principal Investigator — University of Rochester
Locations (1):
- Flaum Eye Institute at the University of Rochester, Rochester, New York, United States